CLINICAL TRIAL: NCT00997230
Title: An NIS Registry for the Epidemiological and Scientific Evaluation of EGFR Mutation Status in Patients With Newly Diagnosed Locally Advanced or Metastatic Non-small Cell Lung Cancer (Stage IIIB/IV Non-small Cell Lung Cancer)
Brief Title: Epidemiological and Scientific Evaluation of EGFR Mutation Status in Patients With Newly Diagnosed Locally Advanced or m
Acronym: REASON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ODE-DUM-2009/1
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Newly Diagnosed Locally Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: EGFR mutation ,newly diagnosed NSCLC, locally advanced or metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is to collect epidemiological data on EGFR mutation status (M+, M-) in a population of predominantly Caucasian ethnicity and to correlate EGFR mutation status with clinico-pathological characteristics (e.g. smoking status, sex, histology, etc). In particular, the study will aim to determine the frequency of EGFR M+ lung cancers in patients with clinico-pathological characteristics that are not commonly associated with EGFR mutation positivity (i.e., smokers, men, and non-adenocarcinoma).

DETAILED DESCRIPTION:
An NIS Registry for the Epidemiological and Scientific evaluation of EGFR mutation status in patients with newly diagnosed locally advanced or metastatic NSCLC (stage IIIB/IV non-small cell lung cancer)

ELIGIBILITY:
Histologically confirmed locally advanced or metastatic NSCLC (stage IIIB/IV). Mixed histology of small cell and non-small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical setting
Sampling Method: Probability Sample
Enrollment: 4243 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to collect epidemiological data on EGFR mutation status (M+, M-) in a population of predominantly Caucasian ethnicity and to correlate EGFR mutation status with clinico-pathological characteristics | Days 1-10

SECONDARY OUTCOMES:
To collect real-life clinical outcome data in all EGFR M+ patients up to and including progression.To collect real-life pharmacoeconomic data (resource use) associated with the diagnosis and treatment of EGFR M+ patients. | Study Days 21-30

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. H. Brasch, Study Director — AstraZeneca Germany; PD Dr. med. Wolfgang Schutte, Principal Investigator — 06120 Halle-Dolau, Germany
Locations (118):
- Germany (118):
  - Research Site, Aachen
  - Research Site, Amberg
  - Research Site, Ansbach
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Berka
  - Research Site, Ballenstedt
  - Research Site, Bamberg
  - Research Site, Bayreuth
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bitterfeld-Wolfen
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Borstel
  - Research Site, Bottrop
  - Research Site, Braunschweig
  - Research Site, Bremen
  - Research Site, Bremerhaven
  - Research Site, Celle
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Cottbus
  - Research Site, Darmstadt
  - Research Site, Deggendorf
  - Research Site, Dessau
  - Research Site, Donaustauf
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Eisenach
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Flensburg
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Freising
  - Research Site, Fulda
  - Research Site, Gerlingen
  - Research Site, Gieben
  - Research Site, Goslar
  - Research Site, Göttingen
  - Research Site, Greifenstein
  - Research Site, Grobhansdorf
  - Research Site, Halle
  - Research Site, Halle-Dolau
  - Research Site, Hamburg
  - Research Site, Hamm
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Hof
  - Research Site, Homburg
  - Research Site, Immenhausen
  - Research Site, Jena
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Koblenz
  - Research Site, Landshut
  - Research Site, Leipzig
  - Research Site, Lemgo
  - Research Site, Leverkusen
  - Research Site, Lostau
  - Research Site, Löwenstein
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Lüneburg
  - Research Site, Lünen
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Minden
  - Research Site, Moers
  - Research Site, Mülheim
  - Research Site, München
  - Research Site, Münnerstadt
  - Research Site, Münster
  - Research Site, Neuss
  - Research Site, Nordhausen
  - Research Site, Northeim
  - Research Site, Nuremberg
  - Research Site, Oberhausen
  - Research Site, Offenbach
  - Research Site, Offenburg
  - Research Site, Oldenburg
  - Research Site, Osnabrück
  - Research Site, Ostfildern
  - Research Site, Paderborn
  - Research Site, Passau
  - Research Site, Querfurt
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Saarbrücken
  - Research Site, Schönebeck
  - Research Site, Solingen
  - Research Site, Sonneberg
  - Research Site, Stralsund
  - Research Site, Stuttgart
  - Research Site, Suhl
  - Research Site, Treuenbrietzen
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Velbert
  - Research Site, Villingen-Schwenningen
  - Research Site, Völklingen
  - Research Site, Wangen/Allgau
  - Research Site, Weiden
  - Research Site, Wiesbaden
  - Research Site, Würselen
  - Research Site, Würzburg
  - Research Site, Zusmarshausen

REFERENCES:
- [Derived] Schuette W, Schirmacher P, Eberhardt WEE, Dietel M, Zirrgiebel U, Muehlenhoff L, Thomas M. Treatment decisions, clinical outcomes, and pharmacoeconomics in the treatment of patients with EGFR mutated stage III/IV NSCLC in Germany: an observational study. BMC Cancer. 2018 Feb 5;18(1):135. doi: 10.1186/s12885-018-4032-3. PMID 29402243